CLINICAL TRIAL: NCT00457704
Title: Carriage and Transmission of Methicillin-Resistant Staphylococcus Aureus (MRSA) in Patients Admitted to Home Care.
Status: Terminated | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Other Study IDs: APHP-SARM-HAD-2003
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Last update posted 2007-04-06 (Estimated); Status verified 2007-04

CONDITIONS: Methicillin-Resistant Staphylococcus Aureus
Keywords: MRSA; Home Care; Risk factors; transmissions; observational study

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Methicillin resistant Staphylococcus aureus (MRSA) which is one of the principal multidrug resistant organisms found in the hospitals all over the world, has recently emerged in the community. However, for the moment (2002), the hospital remains the principal reservoir of MRSA so far and the patients discharged with a MRSA carriage can be the source of MRSA spreading in the community. In particular patients admitted to home care (HC) from acute care facilities represent a patient group with a high risk of MRSA carriage and of being the source of MRSA spreading in the community. The objective of this study is to determine whether HC patients are effectively a MRSA reservoir and a source for MRSA spreading in the community.

For that, from February 2003 to March 2004 any adult patient (except obstetric patient) (approximately 3360 patients for 16 HC settings), will be screened [nasal and skin lesion (if any) swabs] for MRSA carriage within the 48 h before his/her transfer. The patients found to be MRSA carriers will be visited by a physician who will ask patients as well as family members to participate in the study. Each patient and each family member who will have given agreement to participate, will be sampled (nasal swab for both patient and family members, and skin lesion swab for the patients with skin lesions) every month for 12 months by the nurse of the HC setting in which the patient will have been admitted. As soon as the patient will be discharged from HC setting and if the 12 month survey is not finished, patient and family member swab sampling will be performed by the nurse of the research team (NRT) every 3 months until the end of the survey period. These swabs will be transmitted by the NRT to the research center and analyze by the microbial technician of the research center. The bacteriological survey will be accompanied with an epidemiological survey in order to determine the risk factors for a long term MRSA carriage in the patients admitted in HC and also the risk factors for transmitting MRSA to their family.

This multi-centre and multi-investigator study will be performed over a period of 32 months (1 month to prepare the study, 13 months to screen patients with regard to MRSA carriage before their transfer from acute care settings into HC settings, 12 months to survey HC patients and their family members and 6 months to analyze data and prepare publications). Such a study will provide us with descriptive and quantitative data on MRSA strains introduced in the community by HC patients. From the analysis of risk factors of MRSA transmission from these patients to their family members, suggestions to limit this transmission might be drawn.

ELIGIBILITY:
Inclusion Criteria:

* All adults patients positive to MRSA screening at admission in home care and coming from hospital facilities
* All patients MRSA negative leaving in the home of the positive patients
* Written informed consent

Exclusion Criteria:

* Patients admitted in home care for obstetrical or post-partum reasons
* Patients already in the study and being re-hospitalized and re-admitted in home care facilities.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Hélène Nicolas-Chanoine, MD - PHD, Principal Investigator — Assistance Publique des Hôpitaux de Paris - Hôpital Beaujon
Locations (1):
- Dpt Immuno-Microbiologie des Pathologies Infectieuses - Hôpital Beaujon, Clichy, France